CLINICAL TRIAL: NCT05022498
Title: A Replicated Crossover Study Exploring Individual Variability of Postprandial Coronary Heart Disease Risk Markers and Sleep Quality in Response to Acute Exercise in Healthy Young Men
Brief Title: Individual Variability of Coronary Heart Disease Risk Markers and Sleep Responses to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Teesside University (Other)
Responsible Party: Principal Investigator, Professor David Stensel, Professor, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LU-R19-P103
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Coronary Heart Disease; Cardiovascular Risk Factor; Arterial Stiffness; Blood Pressure; Sleep
MeSH Terms: conditions — Coronary Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control 1 (No Intervention): Participants will rest in the laboratory on day 1 and day 2 (08:00-17:00). A high fat breakfast and lunch will be consumed on both days at pre-determined intervals.
- Control 2 (No Intervention): Participants will rest in the laboratory on day 1 and day 2 (08:00-17:00). A high fat breakfast and lunch will be consumed on both days at pre-determined intervals.
- Exercise 1 (Experimental): Participants will complete 60 min of treadmill exercise on day 1 (15:15-16:15). Participants will rest in the laboratory for the remainder of day 1 and throughout day 2 (08:00-17:00). A high fat breakfast and lunch will be consumed on both days at pre-determined intervals.
  Interventions: Behavioral: Exercise
- Exercise 2 (Experimental): Participants will complete 60 min of treadmill exercise on day 1 (15:15-16:15). Participants will rest in the laboratory for the remainder of day 1 and throughout day 2 (08:00-17:00). A high fat breakfast and lunch will be consumed on both days at pre-determined intervals.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 60 min treadmill exercise performed at 60% of maximum oxygen uptake.
  Arms: Exercise 1; Exercise 2

SUMMARY:
The aim of this study is to examine the reproducibility of postprandial coronary heart disease (CHD) risk marker and sleep responses to acute exercise bouts and to quantify the magnitude of individual variability in responses using a replicated crossover design. Healthy, recreationally active men will complete two identical rest control and two identical exercise (60 min at 60% maximum oxygen uptake) conditions in randomised sequences. Fasting and postprandial venous blood samples, arterial blood pressure and arterial stiffness measurements will be taken at pre-determined intervals, and sleep duration and quality will be assessed. Reproducibility and individual variability will be examined using bivariate correlations and linear mixed modelling.

DETAILED DESCRIPTION:
Single bouts of exercise reduce circulating concentrations of postprandial triacylglycerol - an established independent risk marker for coronary heart disease (CHD). The exercise-induced reduction in postprandial triacylglycerol concentrations has been shown to coincide with transient changes in other CHD risk markers, including reductions in postprandial insulin, interleukin-6, arterial stiffness and resting arterial blood pressure, and exercise may also promote sleep duration and quality. Individual variability in these responses is suspected but has not been examined using robust designs and appropriate statistical models. A recent approach to quantify individual variability in the intervention response involves quantifying the participant-by-condition interaction from replicated intervention and comparator arms. Using this approach (the replicated crossover design), the present study will (i) examine whether the postprandial CHD risk marker and sleep responses to acute exercise are reproducible on repeated occasions; and (ii) determine whether there is true individual variability in postprandial CHD risk marker and sleep responses to acute exercise.

A total of 20 healthy, recreationally active men will be recruited. Participants will undertake a preliminary measures visit (visit 1) to confirm eligibility, to undergo anthropometric measurements and to determine maximum oxygen uptake. Participants will complete four, 2-day experimental conditions in randomised sequences separated by at least one week: two identical control and two identical exercise conditions. On day 1 (visits 2, 4, 6 and 8), participants will arrive fasted at 08:00 and a baseline blood sample, blood pressure and arterial stiffness measurement will be taken. Participants will consume a standardised high fat breakfast at 08:45 (0 h) and lunch at 12:45 (4 h). A second arterial stiffness measurement will be taken at 16:45 (8 h). The two control and two exercise conditions will be identical, except that participants will be asked to exercise on the treadmill for 60 minutes at 60% of their maximum oxygen uptake at 15:15 (6.5 h) in both exercise conditions. On day 2 (visits 3, 5, 7 and 9), participants will arrive fasted at 08:00 and will rest in the laboratory throughout the day in the two control and two exercise conditions. Participants will consume a standardised breakfast at 08:45 (0 h) and a standardised lunch at 12:45 (4 h). Venous blood samples will be collected at 0, 0.5, 1, 2, 3, 4, 4.5, 5, 6, 7 and 8 h. Resting arterial blood pressure will be measured at hourly intervals. Arterial stiffness will be measured at 0, 2.5 and 5 h. Sleep duration and quality will be assessed for three nights before and two nights after visits 3, 5, 7 and 9 using a triaxial actigraphy watch.

Reproducibility and individual variability will be explored by correlating the two sets of response differences between exercise and control conditions. Within-participant covariate-adjusted linear mixed models will be used to quantify participant-by-condition interactions. It is hypothesised that (i) control-adjusted postprandial CHD risk marker and sleep responses to acute exercise will be reproducible; and (ii) true interindividual variability will exist in postprandial CHD risk marker and sleep responses to acute exercise beyond any random within-subject variation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45-year-old men;
* Be able to run continuously for 1 hour;
* Body mass index between 18.5 and 29.9 kg/m2;
* No known contradictions to maximal exertion exercise (e.g., recent musculoskeletal injury, congenital heart disease).

Exclusion Criteria:

* Musculoskeletal injury that has affected normal ambulation within the last month;
* Uncontrolled exercise-induced asthma;
* Coagulation or bleeding disorders;
* Heart conditions;
* Diabetes (metabolism will be different to non-diabetics potentially skewing the data);
* Taking any medication that might influence fat metabolism, blood glucose or appetite;
* Smoking (including vaping);
* Dieting or restrained eating behaviours;
* Weight fluctuation greater than 3 kg in the previous 3 months to study enrolment;
* Presence of any diagnosed sleeping disorder;
* A food allergy.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Plasma triacylglycerol concentration | Day 1: fasted; Day 2: fasted (0 hours), 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours and 8 hours
  Fasted plasma triacylglycerol concentration on day 1 and day 2. Time-averaged total area under the curve for triacylglycerol on day 2 in response to exercise and/or feeding.

SECONDARY OUTCOMES:
Plasma glucose concentration | Day 1: fasted; Day 2: fasted (0 hours), 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours and 8 hours
  Fasted plasma glucose concentration on day 1 and day 2. Time-averaged total area under the curve for glucose on day 2 in response to exercise and/or feeding.
Plasma insulin concentration | Day 1: fasted; Day 2: fasted (0 hours), 0.5 hours, 1 hours, 2 hours, 3 hours, 4 hours, 4.5 hours, 5 hours, 6 hours, 7 hours and 8 hours
  Fasted plasma insulin concentration on day 1 and day 2. Time-averaged total area under the curve for insulin on day 2 in response to exercise and/or feeding.
Plasma total cholesterol concentration | Day 1: fasted; Day 2: fasted
  Fasted plasma total cholesterol concentration on day 1 and day 2.
Plasma high-density lipoprotein cholesterol concentration | Day 1: fasted; Day 2: fasted
  Fasted plasma high-density lipoprotein cholesterol concentration on day 1 and day 2.
Plasma low-density lipoprotein cholesterol concentration | Day 1: fasted; Day 2: fasted
  Fasted plasma low-density lipoprotein cholesterol concentration on day 1 and day 2.
Plasma C-reactive protein concentration | Day 1: fasted; Day 2: fasted
  Fasted plasma C-reactive protein concentration on day 1 and day 2.
Apolipoprotein E | Day 1: fasted (baseline)
  Apolipoprotein E genotype at baseline.
Resting arterial blood pressure | Day 1: fasted; Day 2: fasted (0 hours), 1 hours, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours and 8 hours
  Fasted resting systolic and diastolic blood pressure on day 1 and day 2. Time-averaged total area under the curve for systolic and diastolic blood pressure on day 2 in response to exercise and/or feeding.
Resting pulse wave analysis | Day 1: fasted (0 hours), 8 hours; Day 2: fasted (0 hours), 2.5 hours, 5 hours.
  Time-course of resting pulse wave analysis in response to exercise and/or feeding on day 1 and day 2.
Resting pulse wave velocity | Day 1: fasted (0 hours), 8 hours; Day 2: fasted (0 hours), 2.5 hours, 5 hours.
  Time-course of resting pulse wave velocity in response to exercise and/or feeding on day 1 and day 2.
Time in bed | 20 nights (5 nights per condition; three nights before and two nights after visits 3, 5, 7 and 9)
  Total time in bed between 'lights out' to 'lights on'.
Total sleep time | 20 nights (5 nights per condition; three nights before and two nights after visits 3, 5, 7 and 9)
  Total time asleep between 'lights out' to 'lights on'.
Actual wake time | 20 nights (5 nights per condition; three nights before and two nights after visits 3, 5, 7 and 9)
  Total time awake after the first sleep period.
Sleep onset latency | 20 nights (5 nights per condition; three nights before and two nights after visits 3, 5, 7 and 9)
  Total time from 'lights out' to the first sleep epoch.
Sleep efficiency | 20 nights (5 nights per condition; three nights before and two nights after visits 3, 5, 7 and 9)
  Total sleep time expressed as a percentage of time in bed.
Sleep fragmentation index | 20 nights (5 nights per condition; three nights before and two nights after visits 3, 5, 7 and 9)
  Number of times that sleep is terminated after one minute expressed as a percentage of the total sleep time.

CONTACTS AND LOCATIONS:
Overall Officials: David Stensel, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data for all primary and secondary outcome measures will be made available upon request.

REFERENCES:
- [Background] Freese EC, Gist NH, Cureton KJ. Effect of prior exercise on postprandial lipemia: an updated quantitative review. J Appl Physiol (1985). 2014 Jan 1;116(1):67-75. doi: 10.1152/japplphysiol.00623.2013. Epub 2013 Nov 7. PMID 24201708
- [Background] Ashor AW, Lara J, Siervo M, Celis-Morales C, Mathers JC. Effects of exercise modalities on arterial stiffness and wave reflection: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2014 Oct 15;9(10):e110034. doi: 10.1371/journal.pone.0110034. eCollection 2014. PMID 25333969
- [Background] Kredlow MA, Capozzoli MC, Hearon BA, Calkins AW, Otto MW. The effects of physical activity on sleep: a meta-analytic review. J Behav Med. 2015 Jun;38(3):427-49. doi: 10.1007/s10865-015-9617-6. Epub 2015 Jan 18. PMID 25596964
- [Background] Goltz FR, Thackray AE, King JA, Dorling JL, Atkinson G, Stensel DJ. Interindividual Responses of Appetite to Acute Exercise: A Replicated Crossover Study. Med Sci Sports Exerc. 2018 Apr;50(4):758-768. doi: 10.1249/MSS.0000000000001504. PMID 29240652
- [Background] Goltz FR, Thackray AE, Atkinson G, Lolli L, King JA, Dorling JL, Dowejko M, Mastana S, Stensel DJ. True Interindividual Variability Exists in Postprandial Appetite Responses in Healthy Men But Is Not Moderated by the FTO Genotype. J Nutr. 2019 Jul 1;149(7):1159-1169. doi: 10.1093/jn/nxz062. PMID 31132105
- [Background] Atkinson G, Batterham AM. True and false interindividual differences in the physiological response to an intervention. Exp Physiol. 2015 Jun;100(6):577-88. doi: 10.1113/EP085070. Epub 2015 May 13. PMID 25823596
- [Background] Senn S, Rolfe K, Julious SA. Investigating variability in patient response to treatment--a case study from a replicate cross-over study. Stat Methods Med Res. 2011 Dec;20(6):657-66. doi: 10.1177/0962280210379174. Epub 2010 Aug 25. PMID 20739334
- [Background] Senn S. Mastering variation: variance components and personalised medicine. Stat Med. 2016 Mar 30;35(7):966-77. doi: 10.1002/sim.6739. Epub 2015 Sep 28. PMID 26415869
- [Derived] Yang Y, Thackray AE, Shen T, Alotaibi TF, Alanazi TM, Clifford T, Hartescu I, King JA, Roberts MJ, Willis SA, Lolli L, Atkinson G, Stensel DJ. A replicate crossover trial on the interindividual variability of sleep indices in response to acute exercise undertaken by healthy men. Sleep. 2025 Mar 11;48(3):zsae250. doi: 10.1093/sleep/zsae250. PMID 39446630
- [Derived] Shen T, Thackray AE, King JA, Alotaibi TF, Alanazi TM, Willis SA, Roberts MJ, Lolli L, Atkinson G, Stensel DJ. Are There Interindividual Responses of Cardiovascular Disease Risk Markers to Acute Exercise? A Replicate Crossover Trial. Med Sci Sports Exerc. 2024 Jan 1;56(1):63-72. doi: 10.1249/MSS.0000000000003283. Epub 2023 Aug 30. PMID 37703030